CLINICAL TRIAL: NCT01023074
Title: Effects of Training on Central Auditory Function in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B4762-R; NCRAR-VA-04-1205 (Other: Portland VA Medical Center IRB); OHSU - 3188 (Other: Oregon Health Sciences University IRB)
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Multiple Sclerosis
Keywords: MS; CAP
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Non-MS Control (No Intervention): Non-MS control group
- MS: Auditory Training (Active Comparator): MS group receiving auditory training
  Interventions: Behavioral: Auditory training
- MS: Control Activity (Placebo Comparator): MS group not receiving auditory training, doing control activity
  Interventions: Other: MS: Control Activity

INTERVENTIONS:
Behavioral: Auditory training — the study was originally set up so that half of the MS subjects would received auditory training. This intervention has since been discontinued.
  Arms: MS: Auditory Training
Other: MS: Control Activity — MS group not receiving auditory training, doing control activity
  Arms: MS: Control Activity

SUMMARY:
The purpose of this study is to characterize the central auditory processing (CAP) deficits that result from multiple sclerosis (MS).

DETAILED DESCRIPTION:
Five general types of evaluations will be employed over multiple study sessions at the National Center for Rehabilitative Auditory Research (NCRAR). First, a neurologist will review the subject's medical history and perform a neurologic exam to confirm MS diagnosis. Second, peripheral auditory function will be evaluated using a standard set of routine audiometric tests. Additionally, subjects will complete a case history and series of hearing handicap inventories. Third, a battery of behavioral procedures will be used to characterize central auditory processing. Fourth, auditory evoked potential studies will be performed. Emphasis here will be upon evoked potentials whose putative neural generators lie within the central auditory nervous system. Fifth, subjects will receive magnetic resonance imaging (MRI) evaluation to determine sites and amount of neural degeneration.

ELIGIBILITY:
Inclusion Criteria:

* age 21-65 years;
* a clinical or laboratory supported diagnosis of "definite" MS;
* a diagnosis of relapsing-remitting, primary progressive, or secondary progressive MS;
* a Kurtzke Expanded Disability Status Score (EDSS) of 0 to 7.0, inclusive;
* no history of a clinical relapse or change in EDSS for three months preceding entry into the study; and
* a brain MRI scan that shows at least three white-matter lesions on T2-weighted images consistent with MS

Exclusion Criteria:

* current major disease or disorder other than MS (e.g., cancer, end-stage renal disease, end-stage cardiopulmonary disease, post-traumatic stress disorder, diabetes);
* other neurological conditions that could interfere with the ability to respond to tests and questionnaires;
* non-native speaker of English (since test materials are presented in English);
* pregnant (due to potential negative effects on the fetus during fMRI);
* more than a mild degree (less than a 40 dB HL four-frequency pure-tone average [PTA]) of hearing loss bilaterally (since the presence of more than a mild degree of peripheral hearing impairment may impact CAP test results);
* metal implants (due to fMRI constraints); and
* left-handedness

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis N. Bourdette, MD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- MS: Control Activity: MS group not receiving auditory training, doing control activity
  Auditory training: the study was originally set up so that half of the MS subjects would received auditory training. This intervention has since been discontinued.
Period: Overall Study
Arm/Group | Non-MS Control | MS: Auditory Training | MS: Control Activity
Started | 26 | 13 | 13
Completed | 26 | 13 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- MS:Auditory Training: MS group receiving auditory training
  Auditory training: the study was originally set up so that half of the MS subjects would received auditory training. This intervention has since been discontinued.
- Total: Total of all reporting groups
Arm/Group | Non-MS Control | MS:Auditory Training | MS: Control Activity | Total
Number analyzed (Participants) | 26 | 13 | 13 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (12.5) | 52.0 (9.6) | 53.0 (10) | 47.85 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 10 | 35
  Male | 11 | 3 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Electrophysiological Auditory Test
Description: auditory P300 amplitude in response to "rare" 1000 Hz tones
Time Frame: Recordings were conducted during one session
Measure: Mean (Standard Deviation); unit: microvolts
Groups:
- Arm 1: Non-MS control group
- Arm 2: MS group receiving auditory training
  Auditory training: the study was originally set up so that half of the MS subjects would received auditory training. This intervention has since been discontinued.
- Arm 3: MS group not receiving auditory training, doing control activity
  Auditory training: the study was originally set up so that half of the MS subjects would received auditory training. This intervention has since been discontinued.
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 26 | 13 | 13
microvolts | 13.1 (6.7) | 6.4 (4.0) | 6.6 (4.4)

2. Secondary Outcome: Neural Magnetic Resonance Imaging (MRI)
Description: Gray matter volume
Time Frame: Results were recorded during one scanning session
Population: Data reported for 47 study participants who underwent MRI
Measure: Mean (Standard Deviation); unit: cubic cm
Arm/Group | Non-MS Control | MS: Auditory Training | MS: Control Activity
Number analyzed (Participants) | 21 | 13 | 13
cubic cm | 1065 (17) | 990 (22) | 990 (22)

3. Secondary Outcome: SCAN-A: Competing Words Test
Description: The SCAN-A: Competing Words Test assesses participants' auditory processing abilities via a dichotic listening task. Lists of word pairs are presented separately to each ear, and participants repeat the words they hear. Possible range of scores = 0-20, with higher scores indicating better performance.
Time Frame: Test administered during one session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-MS Control | MS: Auditory Training | MS: Control Activity
Number analyzed (Participants) | 26 | 13 | 13
units on a scale | 10.5 (2.2) | 7.5 (3.7) | 7.5 (3.7)

ADVERSE EVENTS:
Arm/Group | Non-MS Control | MS: Auditory Training | MS: Control Activity
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/26 | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No